CLINICAL TRIAL: NCT01745926
Title: Implementation of LUCAS 2 in Helicopter Rescue in South Tyrol
Status: Completed | Type: Observational
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: V/15/11
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CPR: MECHANICAL CHEST COMPRESSION
  Interventions: Device: MECHANICAL CHEST COMPRESSION

INTERVENTIONS:
Device: MECHANICAL CHEST COMPRESSION
  Other Names: LUCAS2

SUMMARY:
Cardiopulmonary resuscitation (CPR) is used to maintain adequate perfusion of vital organs in cardiac arrest patients and is fundamental for the neurological outcome and survival of these individuals. Unfortunately, the quality of CPR may be inadequate due largely to ineffective chest compressions resulting from rescuer fatigue and interruptions in compressions. The LUCAS device (Lund University Cardiopulmonary Assist System, Jolife, Lund, Sweden), introduced in 2002, is the most extensively tested and applied automated alternative to manual CPR for in-hospital care of cardiac arrest patients and during ambulance transfer; the feasibility of application of this device in helicopter emergency medical service (HEMS) operations, however, has never been addressed. The objective of this project is to equip the three active rescue helicopters in South Tyrol with the LUCAS 2 mechanical chest compression device to answer the question: What is the feasibility and efficiency of using this device for prolonged CPR in cardiac arrest patients requiring CPR during HEMS rescue operations and transport?

DETAILED DESCRIPTION:
This is a non-controlled, observational study. Physiological endpoints: MAP (mean arterial pressure); etCO2 (end-tidal expiratory pCO2); ROSC (return of spontaneous circulation); PaO2 (arterial pO2); PaCO2 (arterial pCO2); endpoints to assess feasibility: time from arrival to start of mechanical compressions, problems during transfer into the helicopter and in-field manoeuvers, problems with application of device, problems with patient transfer to hospital premises, hands-off time, personnel requirements.

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest with indication of CPR
* informed consent for those regaining legal competence

Exclusion Criteria:

* declaration of death on site
* contraindications of using the device
* age <18 y

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in cardiac arrest from all causes requiring CPR
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time from arrival of rescue team to start of mechanical compressions | assessed immediatly after the operation is concluded
Presence of abdominal or thoracic lesions caused by automated chest compressor | Assessed at clinical examination during hospital stay (day 1 to day 30) or autopsy

SECONDARY OUTCOMES:
Mean arterial pressure | At hospital arrival (expected between 5 minutes and 1 hour from start CPR)
End-tidal expiratory pCO2 | At hospital arrival (expected between 5 minutes and 1 hour from start CPR)
Return of spontaneous circulation | Could be each moment during CPR
Arterial pO2 | At hospital arrival (expected between 5 minutes and 1 hour from start CPR)
Arterial pCO2 | At hospital arrival (expected between 5 minutes and 1 hour from start CPR)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Brugger, Prof, Study Director — Institute of Mountain Emergency Medicine
Locations (1):
- Eurac research, Bolzano, BZ, Italy